CLINICAL TRIAL: NCT06839482
Title: Efficacy of Robotic Rehabilitation for Neuro Recovery of the Upper Limb in Subacute Stroke Survivors: An International Multicenter Randomized Controlled Trial
Brief Title: Robotic Rehabilitation of the Upper Limb in Subacute Stroke
Acronym: GLORIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 266/IRE/24
Record Dates: First submitted 2025-02-07; First posted 2025-02-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Stroke
Keywords: Stroke; Upper Limb; Hand; Rehabilitation; Robotic- Assisted Therapy; Subacute phase; Activities of Daily Living (ADL); Quality of Life
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In this study all the outcome assessors will be blind to the gruop assignment of the study participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental Group (EG) (Experimental): Participants assigned to Experimental Group (EG) will follow 18+/-3sessions (from a minimum of 3 times to a maximum of 5 times/week) of robotic-assisted treatment for upper limb rehabilitation using the Gloreha Sinfonia (R-Touch Pro; BTL Robotics, USA) robotic device in addition to the standard rehabilitation program.
  Interventions: Device: Robotic Assisted Upper Limb Rehabilitation
- Control Group (CG) (Active Comparator): Participants assigned to Control Group (CG) will follow 18+/-3 sessions (from a minimum of 3 times to a maximum of 5 times/week) of conventional tratment for upper limb rehabilitation in addition to the standard rehabilitation program.
  Interventions: Other: Control Group (CG)

INTERVENTIONS:
Device: Robotic Assisted Upper Limb Rehabilitation — The EG will follow a mixed rehabilitation approach for the upper limb, combining Robotic Assisted Upper Limb Rehabilitation and conventional physical therapy (PT) and/or occupational therapy (OT) with a total daily duration of 90 minutes. The Robotic Assisted UL Rehabilitation's session will last 30 minutes, with the following procedure provided:
  * First week: alternate between passive mobilization exercises, bilateral mode, and therapist-driven mode.
  * Second week: alternate between therapist-driven mode and active-assisted mobilization.
  * Third week: alternate between active-assisted mobilization and active mobilization.
  * Fourth week: alternate between active-assisted mobilization and active mobilization.
  * Fifth week: exclusively perform active mobilization. However, if this proposed progression does not match the patient's motor capabilities, the therapist will optimize the therapeutic program by selecting personalized exercises, following a progressive difficulty approach.
  Other Names: Gloreha Simfonia (R-TOUCH); Robotic treatment for upper limb rehabilitation using the Gloreha Sinfonia (R-Touch)
  Arms: Experimental Group (EG)
Other: Control Group (CG) — The CG will follow a conventional occupational therapy (OT) and physical therapy (PT) program for upper limb rehabilitation, with a total daily duration of 90 minutes. Upper limb rehabilitation exercises will be performed with a therapist who will tailor the treatment according to the patient's clinical characteristics and needs. Specifically, upper limb treatment will consist of motor exercises (shoulder, elbow, wrist, and hand) through a mix of individual sessions with both passive and active interventions where possible.
  Other Names: Conventional treatment for upper limb rehabilitation
  Arms: Control Group (CG)

SUMMARY:
This multicenter international randomized controlled trial (RCT) evaluates the effectiveness of the Gloreha Sinfonia® robotic exoskeleton for upper limb rehabilitation in individuals with subacute post-stroke paresis. The study aims to determine whether robotic-assisted therapy improves voluntary motor control and coordination more effectively than conventional rehabilitation, as measured by the Fugl-Meyer Assessment (FMA) for the upper limb (motor component).

Participants will be randomly assigned to one of two groups:

* Experimental Group (EG): Robotic-assisted upper limb rehabilitation combined with conventional therapy.
* Control Group (CG): Conventional therapy alone including upper limb rehabilitation.

Clinical assessments will be conducted at baseline (T1), post-treatment (T2), and at a 3-month follow-up (T3) using remotely administered scales.

Secondary objectives include evaluating improvements in muscle strength, range of motion, eye-hand coordination, manual dexterity, and functional independence. The study will also assess prognostic factors influencing response to robotic therapy, patient satisfaction, and potential adverse events.

DETAILED DESCRIPTION:
Stroke is a leading cause of disability worldwide, with hemiparesis impairing upper limb function in 75% of affected patients. This deficit significantly reduces patients' independence in activities of daily living (ADLs) and limits social participation. Recovery of upper limb motor function is a primary goal in post-stroke rehabilitation. In recent years, robotic devices for hand rehabilitation have been introduced. The Gloreha Sinfonia® (R-Touch Pro, BTL Robotics) is a robotic exoskeleton that enables repetitive, intensive movements in passive, assisted, and active modes. Despite growing evidence supporting robotics in upper limb rehabilitation, significant gaps remain, including the lack of standardized protocols and the challenge of identifying patient subgroups that would benefit most. This multicenter international RCT aims to address these gaps by evaluating the short- and long-term effectiveness of robot-assisted therapy compared to conventional therapy. The primary objective is to measure the efficacy of robotic rehabilitation using the Fugl-Meyer Motor Assessment (0-66) for the upper limb, a validated scale assessing improvements in strength, active range of motion, eye-hand coordination, and dexterity. This outcome allows for a direct connection between robotic therapy results and motor function, ensuring a precise and replicable evaluation of treatment efficacy relative to conventional therapy. It is hypothesized that robotic treatment with Gloreha Sinfonia R-Touch Pro will significantly improve strength, active range of motion, eye-hand coordination, and manual dexterity, while also promoting autonomy in ADLs and social participation. The study also aims to identify clinical and prognostic factors that influence the response to robotic therapy, assess patient acceptance and satisfaction with the treatment, and monitor for any adverse events. Specifically, secondary objectives of the study are: to assess the impact of robotic treatment on muscle strength, active range of motion, hand-eye coordination, fine motor skills, and dexterity; to examine the effect of treatment on independence in daily living activities and social participation.

Identify clinical characteristics, such as severity of neurological impairment and time from acute event, that best respond to robot-assisted hand therapy; to investigate the influence of treatment initiation timing in relation to the acute event on rehabilitation effectiveness; to assess patient acceptance and satisfaction with the treatment, monitor the occurrence of adverse events, and analyze the effect of treatment on upper limb spasticity. Participants with a stroke diagnosis who meet the inclusion and exclusion criteria will be randomly assigned to one of the following groups: Experimental Group (EG) - robotic treatment for upper limb rehabilitation using the GS robotic device or Control Group (CG) - conventional treatment for upper limb rehabilitation. The study will span 36 months and includes two phases as follows: Phase 1 - Recruitment, baseline evaluations, randomization, rehabilitation intervention, final evaluations, and Phase 2 - Follow-up.

Eligible patients will be randomized into one of two treatment groups (Phase 1): EG or CG. All subjects will be evaluated (Phase 1) with a series of clinical assessments at baseline (T1) and the same assessments will be repeated at the end of the treatment (T2). A 3-month follow-up (Phase 2, T3) will be conducted either through an in-person clinical assessment or a phone interview, based on patient availability, using only remote-administered clinical scales. As for the rehabilitation treatments, the Experimental Group (EG) will receive upper limb rehabilitation assisted by the Gloreha Sinfonia R-Touch Pro device, in addition to conventional therapy, which includes physical therapy (PT) and occupational therapy (OT) and the Control Group (CG) will undergo the same upper limb rehabilitation with only conventional PT and OT treatments, matching the EG's duration for a total of 90 minutes. Both groups will engage in individualized rehabilitation programs, potentially incorporating additional personalized interventions based on each patient's clinical-neurological profile. Randomization will be conducted in a blind manner by an independent collaborator who is not involved in recruitment, intervention, or data collection. Sequentially numbered, opaque, and randomly ordered envelopes containing group assignments will be opened after the initial evaluation, in the participant's presence. Therapists involved will be informed of each patient's group assignment. All data will be collected in compliance with privacy regulations and anonymized on a dedicated platform called RedCAP (Research Electronic Data Capture) https://redcap.sanraffaele.it/. Each center will have access to its own data, with the ability to independently modify and update it. Data will be recorded through the Clinical Report Form (CRF), ensuring systematic and standardized data collection. Descriptive statistical analysis will be performed to adequately represent the clinical and demographic characteristics of the sample, with data presented as frequency (percentage), mean and standard deviation, and median (5th and 95th percentile) for categorical, continuous, and ordinal variables, respectively. Descriptive statistics will ensure score comparability between groups at baseline; an inferential analysis of variables (Kolmogorov-Smirnov test) will be conducted to verify the normality of data distributions. Parametric or non-parametric tests will be applied based on data distribution. The significance level will be set at p<0.05.

In conclusion, the main expected results are: to identify a standardized, reproducible rehabilitation protocol with robotic hand assistance to implement highly customizable rehabilitation protocols; to achieve improved motor recovery in terms of both range of motion and muscle recruitment following upper limb rehabilitation through the Gloreha Sinfonia® (R-Touch Pro) robotic system; to achieve better motor performance following upper limb rehabilitation through the Gloreha Sinfonia® robotic system; to obtain improved eye-hand coordination, manual dexterity, and fine motor skills; to attain greater autonomy in ADL and, consequently, greater participation; to identify any clinical and functional characteristics that impact the rehabilitation outcome with Gloreha Sinfonia R-Touch Pro.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Age 18-90 years
* Paresis of the upper limb following a recent cerebrovascular event (subacute ischemic or hemorrhagic stroke)
* Moderate to mild muscle weakness in the thumb opponens, common finger flexors, and wrist flexors, assessed with complete joint movement in absence of gravity, Medical Research Council Scale (MRC) ≥ 2
* Time from acute event <90 days
* Ability to understand and sign the study informed consent
* Ability to perform study procedures.

Exclusion Criteria:

* Presence of other overlapping neurological disorders
* Presence of osteoarticular or neuromuscular disorders affecting upper limb mobility
* Severe psychiatric disorders
* Severe cognitive (MMSE ≤ 17) and/or language impairment compromising exercise comprehension
* Botulinum toxin injection in the affected upper limb within the last 60 days or planned during the study and follow-up period
* Open wounds, infections, or unprotected skin lesions on the upper limb
* Severe spasticity of the upper limb (biceps and wrist and finger flexors) (MAS > 3)
* Inability to adhere to the exercise program due to low compliance
* Participants who have not signed the informed consent for the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Fugle Meyer Assessment for Upper Limb - Motor Part (score range: 0-66) | Day 0 (T1- basline), day 35 (T2 - After treatment), and day 125 (T3 - 3 months after treatment Follow-Up)
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index designed to evaluate motor function, balance, sensation, and joint integrity in individuals with post-stroke hemiplegia. It is widely used in both clinical and research settings to assess disease severity, track motor recovery, and guide treatment planning.
  In this study, the Motor Part of the FMA for the Upper Limb is the primary outcome measure, with scores ranging from a minimum of 0 to a maximum of 66. A higher score indicates better motor function on the impaired side.

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale (NHISS) | Day 0 (T1- basline), day 35 (T2 - After treatment), and day 125 (T3 - 3 months after treatment Follow-Up)
  The National Institutes of Health Stroke Scale (NIHSS) is a systematic, quantitative assessment tool to measure stroke-related neurological deficit. Its score ranges from 0 to 42, where higher scores indicate greater neurological impairment. In clinical practice it can be used to evaluate and document neurological status in acute stroke patients, determine appropriate treatment and assist in standardizing communication between healthcare practitioners. The NIHSS has been shown to be a predictor of both short and long term outcomes of stroke patients.
Pain scale (NRS 0-10) - at passive mobilization | Day 0 (T1- basline), day 35 (T2 - After treatment), and day 125 (T3 - 3 months after treatment Follow-Up)
  Scores range from 0 to 10, where 0 indicates no pain and 10 represents the worst pain intensity the individual has ever experienced.
Modified Ashworth Scale (MAS) | Day 0 (T1- basline), day 35 (T2 - After treatment), and day 125 (T3 - 3 months after treatment Follow-Up)
  The Modified Ashworth Scale (MAS) is used to assess spasticity. The Modified Ashworth Scale (MAS) has been utilised in the following populations: stroke, spinal cord injury, multiple sclerosis, cerebral palsy, traumatic brain injury, paediatric hypertonia and central nervous system lesions. The test is performed by extending the patients limb's first from a position of maximal possible flexion to maximal possible extension (the point at which the first soft resistance is met). Afterwards, the modified Ashworth scale is assessed while moving from extension to flexion. Scores range from 0 to 4, where 0 indicates no increase in muscle tone and 4 represents a limb that is rigid in flexion or extension.
Medical Research Council Scale (MRC) | Day 0 (T1- basline), day 35 (T2 - After treatment), and day 125 (T3 - 3 months after treatment Follow-Up)
  The Medical Research Council (MRC) Scale for Muscle Strength is a commonly used scale for assessing muscle strength from Grade 5 (normal) to Grade 0 (no visible contraction). The Criteria requires that each of the six muscle groups listed in the table are examined bilaterally, each with a score from 0 to 5 according to the scale in the right hand column.
Box and Block test (BBT) | Day 0 (T1- basline), day 35 (T2 - After treatment), and day 125 (T3 - 3 months after treatment Follow-Up)
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. It can be used with a wide range of populations, including clients with stroke.The BBT is composed of a wooden box divided in two compartments by a partition and 150 blocks. The BBT administration consists of asking the client to move, one by one, the maximum number of blocks from one compartment of a box to another of equal size, within 60 seconds.
Nine Hole Peg Test (NHPT) | Day 0 (T1- basline), day 35 (T2 - After treatment), and day 125 (T3 - 3 months after treatment Follow-Up)
  The Nine-Hole Peg Test (9HPT) is used to measure finger dexterity in patients with various neurological diagnoses. The Nine-Hole Peg Test is administered by asking the client to take the pegs from a container, one by one, and place them into holes on the board as quickly as possible. Participants must then remove the pegs from the holes, one by one, and replace them back into the container.Scores are based on the time taken to complete the activity, recorded in seconds.
Modified Barthel Index (mBI) | Day 0 (T1- basline), day 35 (T2 - After treatment), and day 125 (T3 - 3 months after treatment Follow-Up)
  The modified Barthel Index (mBI) is a well-established patient-centered outcome measure commonly administrated in rehabilitation settings to evaluate the functional status of patients at admission and discharge.
ABILHAND questionnaire | Day 0 (T1- basline), day 35 (T2 - After treatment), and day 125 (T3 - 3 months after treatment Follow-Up)
  The ABILHAND questionnaire is an interview-based, patient-reported measure assessing perceived difficulty in performing manual activities in daily life. It evaluates the active function of the upper limbs and the ability to perform bimanual tasks, regardless of how they are executed. This assessment represents the activity domain of the International Classification of Functioning, Disability, and Health (ICF).
  Validated versions are available for chronic stroke, rheumatoid arthritis, systemic sclerosis, and hand surgery. The scores range from a minimum of 0 to a maximum of 46, with higher scores indicating better performance. All versions, along with assessment details, downloadable materials, and a link to the Rasch analysis, can be accessed through the official website.
Stroke Impact Scale (SIS) | Day 35 (T2 - After treatment), and day 125 (T3 - 3 months after treatment Follow-Up)
  The Stroke Impact Scale (SIS) is a patient-reported outcome measure that evaluates the biopsychosocial aspects of life after stroke. Developed by Duncan et al. at the University of Kansas Medical Center (KUMC) in 1999, it was first published as version 2.0. The original 64-item tool was later refined through Rasch analysis to 59 items, resulting in the current version 3.0. The SIS includes multiple domains, each scored from 0 to 100, with higher scores indicating better function and quality of life. For patients unable to self-report, a proxy version called the Stroke Impact Scale-16 is available.
Robotic Therapy Acceptance Assessment | Day 35 (T2 - After treatment)
  The Robotic Therapy Acceptance Assessment is a questionnaire designed to evaluate patients' perceptions of robotic therapy. It includes items related to various aspects of the experience, namely 'Comfort,' 'Absence of pain,' 'Fatigue,' 'Enjoyment,' 'Advantages,' 'Desire to continue,' and 'Willingness to recommend it to others.' Each item is scored using a Likert scale ranging from 0 to 7, where 0 indicates strong disagreement and 7 represents complete agreement.
Canadian Occupational Performance Measure scale | Day 0 (T1- basline), and day 35 (T2 - After treatment)
  The Canadian Occupational Performance Measure (COPM) is an evidence-based outcome measure designed to assess a client's self-perception of performance in daily activities over time. As a semi-structured interview, it facilitates open dialogue between the client and therapist, focusing on issues most relevant to the client.
  The COPM evaluates two domains: Performance and Satisfaction, both scored on a scale from a minimum of 0 to a maximum of 10. Each domain score represents the mean of 10 items, with each item rated on a Likert scale from 0 to 10. A higher score (10) indicates the best outcome.

OTHER OUTCOMES:
IMU-based targeted Box and Block Test (t-BBT) | Day 0 (T1- basline), and day 35 (T2 - After treatment)
  Instrumental assessment of manual dexterity will be conducted using a sensorized and modified version of the Box and Block Test (BBT). This modified version involves moving 10 cubes from one side of the box to the other positioned on a 5x2 grid. In a subset of EG subjects, kinematic parameters will be measured using Inertial Measurement Units (IMUs), and electrophysiological parameters will be recorded via surface electromyography (sEMG). The assessment will quantify joint kinematics, including range of motion and movement smoothness, as well as upper limb muscle activation patterns, such as muscle onset timing and co-contraction levels. This approach enables a comprehensive evaluation of motor performance during the BBT.

CONTACTS AND LOCATIONS:
Overall Officials: Sanaz Pournajaf, DPT, PhD, Principal Investigator — IRCCS San Raffaele Roma
Locations (20):
- Jefferson Moss-Magee Rehabilitation, Department of PMR, Elkins Park, Pennsylvania, United States
- Czechia (4):
  - Rehabilitation Center of Kladruby, Kladruby
  - Lázně Bělohrad a.s., Centrum komplexní rehabilitace, Lázně Bělohrad
  - Agel Hospital Prostějov, Rehabilitation Centre, Mathonova 1, Clinical Rehabilitation Centre FZV UP, Hněvotínská 3, Olomouc
  - Charles University and General University Hospital in Prague, Prague
- Italy (12):
  - European Society of Physical and Rehabilitation Medicine, SISC in New Technologies and Robotics in Rehabilitation, Rome, Choose One...
  - San Vito Hospital, Rehabilitation Unit, San Vito sullo Ionio, CZ
  - Valduce Hospital, Villa Beretta Rehabilitation Center, Costa Masnaga, LC
  - Department of Rehabilitative Medicine, AUSL Piacenza, Fiorenzuola d'Arda, PC
  - Passignano Hospital, Department of Specialized Medicine, Usl Umbria 1, Passignano sul Trasimeno, Perugia
  - Fondazione Policlinico Universitario Campus Bio-Medico di Roma, UOC di Medicina Fisica e Riabilitativa-CESA, Rome, RM
  - IRCCS San Raffaele Roma, Rome, RM
  - ASST Papa Giovanni XXIII, Bergamo
  - University of Catanzaro "Magna Graecia", Catanzaro
  - IRCCS Fondazione Don Gnocchi, Florence
  - Riuniti Hospital, Neurorehabilitation, Spinal Cord Rehab. and Functional Recovery Section, Foggia
  - IRCCS Centro Neurolesi Bonino-Pulejo, Innovation Technology Laboratory, Messina
- Medical Centre for Rehabilitation Treatment "Consilium", Moscow, Russia
- Centro Lescer, Occupational Therapy and Physical Therapy Department, Madrid, Spain
- Chiang Mai University, Department of Occupational Therapy, Faculty of Associated Medical Sciences, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared with qualified researchers upon reasonable request, following ethical and regulatory approvals.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual participant data (IPD) will be available upon publication of the main results and will remain accessible for at least five years.
Access Criteria: Qualified researchers may request access to the data by submitting a proposal outlining their research objectives. Access will be granted upon ethical and regulatory approval and under a data-sharing agreement.

REFERENCES:
- See also: 2015 American Heart Association/American Stroke Association Focused Update of the 2013 Guidelines for the Early Management of Patients With Acute Ischemic Stroke Regarding Endovascular Treatment: A Guideline for Healthcare Professionals From the American — http://pubmed.ncbi.nlm.nih.gov/26123479/
- See also: S.P. and E.A. Diffusion, "Ictus cerebrale: SPREAD linee guida italiane," 2016. — http://isa-aii.com/linee-guida-spread-viii-edizione/
- See also: C.J. Winstein et al., "Guidelines for Adult Stroke Rehabilitation and Recovery: A Guideline for Healthcare Professionals from the American Heart Association/American Stroke Association," Stroke, 47(6), 2016. — http://pubmed.ncbi.nlm.nih.gov/27145936/
- See also: Evidence-based review of stroke rehabilitation, 20th Edition (EBRS) — http://www.ebrsr.com/evidence-review
- See also: Task-Based Mirror Therapy Augmenting Motor Recovery in Poststroke Hemiparesis: A Randomized Controlled Trial — http://pubmed.ncbi.nlm.nih.gov/26096318/
- See also: Mirror Therapy for Stroke Rehabilitation — http://pubmed.ncbi.nlm.nih.gov/26723854/
- See also: Clinical relevance of action observation in upper-limb stroke rehabilitation: a possible role in recovery of functional dexterity. — http://pubmed.ncbi.nlm.nih.gov/22235059/
- See also: Motor impairment as a predictor of functional recovery and guide to rehabilitation treatment after stroke — https://pubmed.ncbi.nlm.nih.gov/11944745/
- See also: Action Observation Therapy — http://pubmed.ncbi.nlm.nih.gov/17499164/
- See also: Use of the Medical Research Council Muscle Strength GradingSystem in the Upper Extremity — https://pubmed.ncbi.nlm.nih.gov/17275587/
- See also: Electromechanical and robot-assisted arm training for improving activities of daily living, arm function, and arm muscle strength after stroke. — http://pubmed.ncbi.nlm.nih.gov/30175845/
- See also: Probability of regaining dexterity in the flaccid upper limb: impact of severity of paresis and time since onset in acute stroke. — https://pubmed.ncbi.nlm.nih.gov/12907818/
- See also: Upper limb robot-assisted rehabilitation versus physical therapy on subacute stroke patients: A follow-up study. — https://pubmed.ncbi.nlm.nih.gov/31987544/
- See also: Reliability of the Fugl-Meyer assessment for testing motor performance in patients following stroke. — https://pubmed.ncbi.nlm.nih.gov/8316578/
- See also: Reliability and validity of the Medical Research Council (MRC) scale and a modified scale for testing muscle strength in patients with radial palsy. — https://pubmed.ncbi.nlm.nih.gov/19020701/
- See also: Stroke Scale — https://strokengine.ca/en/assessments/nihss/
- See also: The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. — https://pubmed.ncbi.nlm.nih.gov/1135616/
- See also: Modified Ashworth Scale. [Updated 2023 May 1]. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing — http://www.ncbi.nlm.nih.gov/books/NBK554572/
- See also: Adult norms for the Box and Block Test of manual dexterity — https://pubmed.ncbi.nlm.nih.gov/3160243/
- See also: Hand strength and dexterity — https://pubmed.ncbi.nlm.nih.gov/5551515/
- See also: abilhand — http://rssandbox.iescagilly.be/abilhand.html
- See also: Rasch analysis of a new stroke-specific outcome scale: The Stroke Impact Scale. — https://pubmed.ncbi.nlm.nih.gov/12881816/
- See also: Acceptability of robotic technology in neuro-rehabilitation: preliminary results on chronic stroke patients. — https://pubmed.ncbi.nlm.nih.gov/24461799/